CLINICAL TRIAL: NCT06237218
Title: Effets du Programme COTID (Community Occupational Therapist in Dementia) et d'Une Prise en Soins ergothérapique Habituelle Sur la récidive de Chutes à 12 Mois de Personnes âgées Atteintes de Troubles Neurocognitifs et Ayant été hospitalisées Pour Chute, après Leur Retour à Domicile
Brief Title: Effects of the COTID (Community Occupational Therapist in Dementia) Program and Usual Occupational Therapy Care on Recurrence of Falls at 12 Months in Elderly People With Neurocognitive Disorders Who Had Been Hospitalized for Falls, After Their Return Home
Acronym: ErgoFalls
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 87RI21_0009_ErgoFallsPilote
Record Dates: First submitted 2023-10-26; First posted 2024-02-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Nervous System Diseases
Keywords: Dementia
MeSH Terms: conditions — Nervous System Diseases; Dementia

STUDY DESIGN:
Intervention Model Description: Double-blind randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COTID program (Experimental): The intervention takes place entirely in the homes of elderly people with neurocognitive disorders.
  It takes an average of 10 hours of intervention per treatment, spread over 5 to 10 weeks.
  The COTID program is divided into several phases:
  * Phase A: Problem definition and analysis
  * Phase B: Formulation of objectives and treatment plan
  * Phase C: Implementation of the treatment plan.
  Interventions: Behavioral: COTID program
- Routine care (No Intervention): Patient's needs without a COTID program.

INTERVENTIONS:
Behavioral: COTID program — COTID is a support program for people with Alzheimer's disease, designed to help them remain at home, including their primary caregiver.
  Arms: COTID program

SUMMARY:
This project will enable optimization of specific carried out by occupationist for older adults discharged from hospital for falls:

* on the environmental dimension at the participant's home
* on the involvement of the caregiver since they are also involved in the care of the patient
* on the recurrence of falls and rehospitalizations in order to improve the quality of life by reassuring the elderly person when traveling
* on limiting loss of autonomy and staying at home. The occupational therapist will entrust the caregiver with a support role. The participant will feel more involved in the participant's care (thus reducing the feeling of helplessness). His actions will allow him to strengthen his sense of competence and will prevent him from physical and psychological exhaustion.

DETAILED DESCRIPTION:
Falls constitute the greatest cause of loss of autonomy among people aged over 65 and are often the cause of injuries leading to hospitalization and therefore significant costs. Additionally, people who have fallen before are at greater risk of falling again. People aged 65 and over with dementia fall 3 times more than people without the condition. The physical and psychological consequences of these falls in patients with dementia accelerate their loss of autonomy and ultimately lead to admission to an institution.

Occupational therapy assessment in the patient's home is an effective approach to reducing falls in the general population. Indeed, the occupational therapist's care consists of carrying out a complete assessment to highlight the links that exist between a person and their abilities, their occupations in the broad sense and the environment in which their occupations take place. The occupational therapist then proposes a personalized intervention plan (objectives and means) and follow-up which may consist of the installation of technical and technological aids, home design, advice and information for people and their caregivers.

The COTID (Community Occupational Therapist in Dementia) program is a tool for describing the stages of an occupational therapy program based on evidence (scenario-based), according to a systemic approach focused on older people with dementia and their caregivers. This has been validated and widely used in the Netherlands since 2009. Indeed, it has shown its effectiveness in terms of successfully keeping elderly people with dementia at home but also in preventing the risk of caregiver burnout. through systemic care for the couple.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 75 years old
* Living at home (excluding nursing home or long-term care facilities)
* Hospitalized for fall
* Presenting major mild to moderate dementia (MMSE > 16)
* Accompanied by a caregiver with sufficient presence to meet study procedures: at investigator's discretion at the investigator's discretion
* Having given free, informed and written consent signed by the patient
* Whose caregiver has given free, informed consent written and signed by him/herself
* Affiliated or beneficiary of social security

Exclusion Criteria:

* With serious, life-threatening pathology(ies) or in palliative care
* Participating in an educational fall program on the theme of falls, run by an occupational therapist by an occupational therapist
* Receiving regular occupational therapy treatment on the day of inclusion (day care daily hospitalization)
* Participating in a clinical research protocol have an impact on the occurrence of a fall (at the investigator's discretion)
* Not matching with the fall definition from Kellogg's definition of a fall (loss of consciousness, sudden onset of paralysis paralysis or epileptic seizure)
* Presenting a very significant post-fall syndrome:

score of 4/4 on the "Get-up early" questionnaire

* unable to read or write
* Participant under legal guardianship (curator, guardian, legal protector)
* Dementia with rapid neurocognitive degeneration degeneration with frontal and language impairment (at the investigator's discretion).

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2027-03-08 (Estimated)

PRIMARY OUTCOMES:
Assessing the impact of the COTID program | 12 months
  Reference will be falls recurrence

SECONDARY OUTCOMES:
Recurrent falls | 12 months
  The cumulative incidence of new falls between the two groups
Rehospitalization | 12 months
  The rehospitalization rate
Institutional admissions | 12 months
  The rate of institutional admissions
Loss of functional autonomy | 12 months
  Scores: Activities of Daily Living, Instrumental Activities of Daily Living
Functional autonomy | 12 months
  Scores: Activities of Daily Living, Occupational efficiency
Fragility profile | 12 months
  Fragility according to Fried criteria
The caregiver's burden | 12 months
  Zarit score comparison between the 2 arms
Coping strategies for caregivers | 12 months
  According to the Ways of Coping Checklist
Learning retention | Between months 6 and months 12
  According to the Ways of Coping Checklist

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No